CLINICAL TRIAL: NCT05395728
Title: Relationship Between Deflating the Tracheostomy Tube Cuff During Wean Mechanical Ventilation and Time for Decannulation
Brief Title: Deflating the Tracheostomy Tube Cuff and Time for Decannulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Principal Investigator, Cassiano Teixeira, Principal Investigator, Hospital Moinhos de Vento
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Tracheostomy tube cuff
Record Dates: First submitted 2022-05-15; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Deglutition Disorders; Tracheostomy Complication
Keywords: deglutition disorders; Tracheostomy
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial. Group 1: deflate the cuff at the beginning of the weaning protocol from mechanical ventilation.
  Group 2: deflate after complete weaning from mechanical ventilation.
Who Masked: Investigator
Masking Description: A single person blinded in the study will draw the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Deflate the cuff at the beginning of the mechanical ventilation weaning protocol
  Interventions: Other: Deflate the tracheostomy cuff early
- Group 2 (Active Comparator): Deflate the cuff after complete weaning from mechanical ventilation
  Interventions: Other: Deflate the tracheostomy cuff after complete weaning mechanical ventilation

INTERVENTIONS:
Other: Deflate the tracheostomy cuff early — The tracheostomy cuff will be early deflated, on beginning the weaning mechanical ventilation
  Arms: Group 1
Other: Deflate the tracheostomy cuff after complete weaning mechanical ventilation — The tracheostomy cuff will be deflated onl twenty four hours after complete weaning mechanical ventilation
  Arms: Group 2

SUMMARY:
Introduction: Inpatients in an intensive care unit can need tracheostomy. To start the tracheostomy decannulation process, one of the procedures is to deflate the cuff. Purpose: Check whether to set the cuff early reduction of tracheostomy use. Methodology: This is a randomized clinical trial, where the cuff of the experimental group will be deflated from the beginning of periods without mechanical ventilation, and the control group after 24 hours without mechanical ventilation. Will be included tracheostomized patients weaning the mechanical ventilation, and excluded those who do not have the consent form signed.

DETAILED DESCRIPTION:
The general objective is to verify that patients who go through the process of deflating the cuff from the initiation of weaning from mechanical ventilation meet criteria for decannulation before patients who deflate the cuff only after 24 hours of weaning.

The study will be carried out in the Intensive Care Unit of Hospital Moinhos de Vento, located in the city of Porto Alegre/RS

The evaluation must take place according to the following steps, after the request of the medical team: Check if the patient meets the inclusion criteria; Raffle to verify if the patient will participate in the study group or the group control; The draw will be performed by a person blinded to the study; Application of the informed consent to the patient or legal guardian; Collection of data in medical records; Explain the procedures to the patient; Position the patient as seated as possible; Tracheal aspiration; Deflate the cuff; Tracheal aspiration after deflating the cuff; Collect data from the moment of the evaluation; The assessment will be recorded in the patient's electronic medical record by the speech therapist at the service; Monitor the moment the patient reaches the criteria for decannulation after complete weaning from mechanical ventilation. For the control group, the same procedures will be performed after complete 24 continuous hours without the use of mechanical ventilation

The following clinical data will be collected in electronic medical records: sex, date of birth, age, reason for hospitalization, comorbidities, date of hospitalization, date of orotracheal intubation procedure and date of tracheostomy procedure. At the time of evaluation, the following variables will be collected: tracheostomy; time in ayre (without mechanical ventilation); oxygen saturation, heart and respiratory rate before and after cuff deflation; cough strength (weak, strong, absent); cough quality (effective, ineffective); saliva swallowing (spontaneous, on command, absent), date of decannulation.

After the evaluation, the following variables will be collected to consider the patient decannulation: permeability of the air passage during occlusion of the tracheostomy, tolerance of occluded tracheostomy, management of secretion and efficiency of saliva swallowing.

ELIGIBILITY:
Inclusion Criteria:

* Request for speech therapy evaluation by the medical team
* Use of tracheostomy
* Indication to start the weaning process from mechanical ventilation
* Consent to the Free and Informed Consent Form by the patient or by the legal responsible

Exclusion Criteria:

- Diagnosis of head and neck cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-12 (Estimated)

PRIMARY OUTCOMES:
Time to reach decannulation | Will be measured in days. Two points will be considered: day that the cuff was deflated and day of decannulation, with an estimated period of 4 weeks.
  The time between deflating the cuff for the first time and the day of decannulation will be counted for the both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Cassiano Teixeira, Study Director — Hospital Moinhos de Vento; Hellen Antunes, Principal Investigator — Hospital Moinhos de Vento
Locations (1):
- Hellen de Araujo Antunes, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
The data will be disclosed in a general way, only distributed in groups. Individual data of research participants will not be disclosed.

REFERENCES:
- [Background] CALLON J, LAMONT C, DYSON S, et al. Early cuff deflation in tracheostomised patients requiring ventilatory support. Critical Care, v. 23, 2019.